CLINICAL TRIAL: NCT06103695
Title: Open Label, Observational Study, Evaluating VTAMA® (Tapinarof) Cream, 1% QD in Psoriasis Patients Being Treated With Biologic Agents.
Brief Title: Vtama in Psoriasis Patients Being Treated With Biologics.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Psoriasis Treatment Center of Central New Jersey (Other)
Responsible Party: Principal Investigator, Jerry Bagel, MD, MS, Psoriasis Treatment Center of Central New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC10
Record Dates: First submitted 2023-10-19; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — tapinarof

STUDY DESIGN:
Intervention Model Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vtama (Other): open label Vtama
  Interventions: Drug: Tapinarof

INTERVENTIONS:
Drug: Tapinarof — Add on Vtama (tapinarof) to biololgic therapy

SUMMARY:
Open label study to assess 12 weeks of add-on VTAMA® (tapinarof) Cream, 1% QD in patients with ≥3% BSA who have received biologic therapy for at least 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult ≥ 18 years of age;
2. Diagnosis of chronic plaque-type
3. Patient with ≥3% BSA
4. Patient has been treated with biologic for a minimum of 24 weeks
5. Able and willing to give written informed consent prior to performance of any study-related procedures.

Exclusion Criteria:

1. ≤3% BSA
2. Patient not receiving biologic agent, or receiving biologic agent <24weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Body surface area ≤1% | 12 weeks
  Patients who achieve body surface area of ≤1%

CONTACTS AND LOCATIONS:
Locations (1):
- Schweiger Derm Group, East Windsor, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No